CLINICAL TRIAL: NCT05280327
Title: The Effect of Virtual Reality Applications in Travail on Perceived Labor Pain and Satisfaction in Primiparous: A Design Based Study
Brief Title: Virtual Reality Effect on Labor Pain and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, zeliha sunay, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/603
Record Dates: First submitted 2021-12-27; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Satisfaction; Labor Pain
Keywords: Primiparous; Birth Pain; Birth Satisfaction; Virtual Reality; Midwifery
MeSH Terms: conditions — Personal Satisfaction; Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): virtual reality application
  Interventions: Other: Virtual Reality Application
- control group (No Intervention): standard care group

INTERVENTIONS:
Other: Virtual Reality Application — The pregnant women in the experimental group were played by the researcher during the active and transitional phases of labor with virtual reality glasses, which were designed for research and included methods used to cope with labor pain
  Arms: experimental group

SUMMARY:
The primiparous women wore virtual glasses during labor, playing games and exercising. pregnant women were divided into two groups. Experimental and control groups each consisted of 60 pregnant women.

DETAILED DESCRIPTION:
Aim: The research was carried out to determine the effect of virtual reality application in labor on perceived labor pain and satisfaction levels in primiparous.

Material and Method: The study was conducted in a randomized controlled manner with a total of 120 primiparous women who applied to the delivery room of Elazig Fethi Sekin City Hospital between June 2020 and June 2021 (60 Experiments, 60 Controls). The pregnant women in the experimental group were played by the researcher during the active and transitional phases of labor with virtual reality glasses, which were designed for research and included methods used to cope with labor pain. Except for routine care, no application was made to the pregnant women in the control group. In order to determine the pain level of the pregnant women, SDS and SCS were applied four times, before and after the Virtual Reality applications. After delivery, DME-C was applied to both groups.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women who were able to communicate verbally
* Between 37-42 weeks of pregnancy
* Single, live fetus and head presentation
* Cervical opening <4 cm based on the labor follow-up form at admission to the delivery room, were included in the sample

Exclusion Criteria:

* Women with a risky pregnancy diagnosis (such as preeclampsia, placenta previa, gestational diabetes)
* Obstetric complications in labor (such as fetal distress, bleeding)
* Visual and hearing problems
* Any pharmacological pain-reducing method applied, were excluded from the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
change in pain score within one hour during the latent phase | SDS was applied as a pre-test to all pregnant women in both groups in the latent phase. One hour later, it was applied to all pregnant women in both groups as a post-test.
  In order to determine the pain level of the pregnant women, SDS was applied four times, before and after the Virtual Reality applications in the latent and active phases. SDS is rated from Scale 0 (zero) to 10 (ten). In the scale, 0 (zero) means no pain, 10 (ten) means unbearable pain. The person can mark according to the severity of the pain on this scale.
change in pain score within one hour during the the active phase | SDS was applied as a pre-test to all pregnant women in both groups in the active phase. One hour later, it was applied to all pregnant women in both groups as a post-test.
  In order to determine the pain level of the pregnant women, SDS was applied four times, before and after the Virtual Reality applications in the latent and active phases. SDS is rated from Scale 0 (zero) to 10 (ten). In the scale, 0 (zero) means no pain, 10 (ten) means unbearable pain. The person can mark according to the severity of the pain on this scale.
change in pain score within one hour during the latent phase | SCS was applied as a pre-test to all pregnant women in both groups in the latent phase. One hour later, it was applied to all pregnant women in both groups as a post-test.
  In order to determine the pain level of the pregnant women, SCS was applied four times, before and after the Virtual Reality applications in the latent and active phases. This scale is based on the person choosing the most appropriate word to describe the pain condition. Pain intensity ranges from mild to unbearable. The severity of pain is defined in five categories and is scored as (1) "mild", (2) "disturbing", (3) "severe", (4) "very severe", and (5) "unbearable". The advantages of the scale are that it is easy to apply and simple to classify.
change in pain score within one hour during the the active phase | SCS was applied as a pre-test to all pregnant women in both groups in the active phase. One hour later, it was applied to all pregnant women in both groups as a post-test.
  In order to determine the pain level of the pregnant women, SCS was applied four times, before and after the Virtual Reality applications in the latent and active phases. This scale is based on the person choosing the most appropriate word to describe the pain condition. Pain intensity ranges from mild to unbearable. The severity of pain is defined in five categories and is scored as (1) "mild", (2) "disturbing", (3) "severe", (4) "very severe", and (5) "unbearable". The advantages of the scale are that it is easy to apply and simple to classify.

CONTACTS AND LOCATIONS:
Overall Officials: zeliha sunay, Phd, Principal Investigator — munzur üniversitesi
Locations (1):
- İnönü University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
we don't share individual participant data with other researchers

REFERENCES:
- [Result] Gur EY, Apay SE. The effect of cognitive behavioral techniques using virtual reality on birth pain: a randomized controlled trial. Midwifery. 2020 Dec;91:102856. doi: 10.1016/j.midw.2020.102856. Epub 2020 Sep 28. PMID 33478718